CLINICAL TRIAL: NCT01658306
Title: A Random Controlled, Double-Blind Clinical Trial: Remote Ischemic Preconditioning and Cerebral Small Vessel Disease
Brief Title: Clinical Trial on Remote Ischemic Preconditioning and Cerebral Small Vessel Disease
Acronym: RIPC-SVD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Ji Xunming, Professor of Neurosurgery, Vice-President of Xuan Wu Hospital, Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D111107003111008
Record Dates: First submitted 2012-07-26; First posted 2012-08-07 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Cerebral Small Vessel Disease
Keywords: remote ischemic preconditioning; random-controlled; double blind; RIPC
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- remote ischemic preconditioning (Experimental): Receiving remote ischemic preconditioning (RIPC) treatment with pressure set at 200 mmHg.
  Interventions: Procedure: remote ischemic preconditioning
- placebo remote ischemic preconditioning (Sham Comparator): Receiving sham RIPC treatment with pressure set at 50 mmHg
  Interventions: Procedure: sham remote ischemic preconditioning

INTERVENTIONS:
Procedure: remote ischemic preconditioning — RIPC consists of five 5-min cycles of right upper arm ischemia/reperfusion, induced by an automated cuff-inflator placed on the right upper arm which is inflated to 200 mmHg for 5mins followed by deflating the cuff for 5mins, each patient in the RIPC group will have the treatment twice a day for two weeks.
  Arms: remote ischemic preconditioning
Procedure: sham remote ischemic preconditioning — Sham RIPC consists of five 5-min cycles of right upper arm ischemia/reperfusion, induced by an automated cuff-inflator placed on the right upper arm which is inflated to 50 mmHg for 5mins followed by deflating the cuff for 5mins, each patient in the placebo RIPC group will have the treatment twice a day for two weeks.
  Arms: placebo remote ischemic preconditioning

SUMMARY:
The hypothesis of this study is that remote ischemic preconditioning (RIPC) might have a beneficial effect on outcomes of cerebral small vessel disease (CSV).

DETAILED DESCRIPTION:
CSV constitutes an important type of ischemic stroke due to a generalized hypo-perfusion of brain. Few treatment methods are available except some beneficial effect shown with nimodipine. The potential treatment effect of RIPC on protection of brain from cerebral small vessel disease has not been investigated. The investigators designed this randomized, double-blind, controlled clinical trial to examine (1) whether RIPC has a beneficial effect on brain lesions of CSV, and (2) whether RIPC can protect patients of CSV from cognitive deterioration. There are 2 arms in this trial: One arm is RIPC treatment, the other one is sham RIPC treatment. Brain lesions will be quantified by volumetric MRI, and Xe-CT will be used to evaluate cerebral blood perfusion. Cognitive function will be evaluated by mini-mental state examination (MMSE) and the Montreal Cognitive Assessment (MoCA).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 40-80 years;
2. Ischemic cerebrovascular event onset, if any, must be within 6 months;
3. TCD and carotid ultrasound exclude vascular narrow that can cause hemodynamic changes (usually >50% narrow lumen);
4. MRI confirmed the presence of lacunar infarction and / or generalized white matter lesions;
5. Written consent was obtained from the subject.

Exclusion Criteria:

1. History of intracranial hemorrhage;
2. Significant bleeding from other parts of the body;
3. History of atrial fibrillation;
4. History of myocardial infarction within six months;
5. Moyamoya disease or vasculitis;
6. Hereditary small vessel disorders, such as CADASIL, FABRY, and mitochondrial encephalo-myopathy;
7. Significant bleeding-coagulation dysfunction;
8. Abnormal blood pressure, glucose and/or lipids after restrict treatment regimen;
9. Severe liver/kidney disease, cancer or critical illness of internal medicine and surgery.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
changes in brain lesions | 0-24 months
  Volumetric MRI will be used for calculating changes in the number of lacunar infarctions and the total volume of white matter lesions

SECONDARY OUTCOMES:
Changes in the cognitive function | 0-24 months
  Cognitive function will be evaluated by mini-mental state examination (MMSE) and the Montreal Cognitive Assessment (MoCA).
Changes in the cerebral blood perfusion | 0-24 months
  Cerebral blood perfusion will be evaluated by Xe-CT.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, M.D., Ph.D., Principal Investigator — Xuan Wu Hospital of Capital Medical University
Locations (1):
- Xuan Wu Hospital, Beijing, China

REFERENCES:
- [Derived] Wang Y, Meng R, Song H, Liu G, Hua Y, Cui D, Zheng L, Feng W, Liebeskind DS, Fisher M, Ji X. Remote Ischemic Conditioning May Improve Outcomes of Patients With Cerebral Small-Vessel Disease. Stroke. 2017 Nov;48(11):3064-3072. doi: 10.1161/STROKEAHA.117.017691. Epub 2017 Oct 17. PMID 29042490
- [Derived] Mi T, Yu F, Ji X, Sun Y, Qu D. The Interventional Effect of Remote Ischemic Preconditioning on Cerebral Small Vessel Disease: A Pilot Randomized Clinical Trial. Eur Neurol. 2016;76(1-2):28-34. doi: 10.1159/000447536. Epub 2016 Jun 29. PMID 27351719